CLINICAL TRIAL: NCT05283863
Title: Direct Comparison of Spinal Cord Stimulator Parameter Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-13-29
Record Dates: First submitted 2021-12-23; First posted 2022-03-17 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Stimulation; High-frequency Stimulation; High-density Stimulation

STUDY DESIGN:
Intervention Model Description: All subjects underwent two weeks of conventional stimulation, followed by randomization to receive either subthreshold high-density (HD) or sham stimulation; this was followed by a crossover during which the participants who had received subthreshold HD stimulation were treated with sham and vice versa.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-Frequency Stimulation, Then Placebo Stimulation (Experimental): Participants first receive sub-threshold high-frequency spinal cord stimulation (1200 Hz frequency, 200 μsec pulse width, and an amplitude 90% of the threshold for detection of a sensory percept) for 2 weeks. After a 2-week washout period, they then receive sham spinal cord stimulation (1200 Hz at 0 V amplitude) for 2 weeks.
  Interventions: Device: High-frequency stimulation; Device: Sham Stimulation
- Placebo Stimulation, Then High-Frequency Stimulation (Sham Comparator): Participants first receive sham spinal cord stimulation (1200 Hz at 0 V amplitude) for 2 weeks. After a 2-week washout period, they then receive sub-threshold high-frequency spinal cord stimulation (1200 Hz frequency, 200 μsec pulse width, and an amplitude 90% of the threshold for detection of a sensory percept) for 2 weeks.
  Interventions: Device: High-frequency stimulation; Device: Sham Stimulation

INTERVENTIONS:
Device: High-frequency stimulation — Patients in this group will receive sub-threshold high-frequency (aka 1200Hz) spinal cord stimulation for 2 weeks.
Device: Sham Stimulation — Patients in this group will receive receive sham spinal cord stimulation (aka no stimulation) for 2 weeks.

SUMMARY:
(Primary)

1. To compare the clinical effects and side effects of two different stimulation strategies that do not produce any sensory percept (1000 Hz and placebo) on clinical benefit for electrodes implanted for chronic pain as measured by the Visual Analog Pain Scale for back and leg pain, the Brief Pain Inventory, the 36-Item Short Form Survey (SF-36), and the Pain Vigilance and Awareness Questionnaire.

   (Secondary)
2. To compare the clinical effects of the subthreshold (paresthesia-free) stimulation patterns with conventional (paresthesia-producing) stimulation patterns to evaluate the necessity of paresthesias and current amplitudes on clinical benefit for pain.
3. To identify the ability of subthreshold high-frequency to improve axial pain or the affective component of pain.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind study of different stimulation patterns in patients undergoing implantation of neurostimulator systems for chronic medically intractable neuropathic pain. Research participants will be individuals who have undergone implantation of neurostimulator electrodes into the spinal column or peripheral nervous system for clinical treatment of neuropathic pain. All patients will already have undergone empiric programming of the stimulator using conventional settings (typically 40-60 Hz, 350-450 usec pulse width). However, other stimulation parameters, including high-frequency stimulation, are also feasible and FDA-approved using the implanted device, and it is possible to do this without producing a sensory percept, which makes it possible to test efficacy in a double blind manner. For this study, two different stimulation parameters will be tested during four two-week periods: 1000 Hz and placebo. Clinical response and side effect profile for each setting will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Diagnosis of chronic neuropathic pain for which placement of electrodes into the spinal column is planned for clinical indications (failed back surgery syndrome, peripheral neuropathy or complex regional pain syndrome)
* History of implantation of spinal cord stimulation system with rechargeable implanted neurostimulator

Exclusion Criteria:

* Significant dementia or other condition preventing informed consent by the patient.
* Current drug or alcohol abuse or dependence.
* Uncontrolled depression or anxiety or failure to pass psychological screening for spinal cord stimulation.
* Inability or unwillingness to cooperate with clinical testing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Sweet, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Sweet J, Badjatiya A, Tan D, Miller J. Paresthesia-Free High-Density Spinal Cord Stimulation for Postlaminectomy Syndrome in a Prescreened Population: A Prospective Case Series. Neuromodulation. 2016 Apr;19(3):260-7. doi: 10.1111/ner.12357. Epub 2015 Oct 20. PMID 26481726

RESULTS

PARTICIPANT FLOW:
Groups:
- High-Frequency Stimulation, Then Placebo Stimulation: Participants first received sub-threshold high-frequency spinal cord stimulation (1200 Hz frequency, 200 μsec pulse width, and an amplitude 90% of the threshold for detection of a sensory percept) for 2 weeks. After a 2-week washout period, they then received sham spinal cord stimulation (1200 Hz at 0 V amplitude) for 2 weeks.
Period: First Intervention (14 Days)
Arm/Group | High-Frequency Stimulation, Then Placebo Stimulation | Placebo Stimulation, Then High-Frequency Stimulation
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | High-Frequency Stimulation, Then Placebo Stimulation | Placebo Stimulation, Then High-Frequency Stimulation
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Second Intervention (14 Days)
Arm/Group | High-Frequency Stimulation, Then Placebo Stimulation | Placebo Stimulation, Then High-Frequency Stimulation
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were randomized to the conventional spinal cord stimulation group
Groups:
- High-Frequency Stimulation, Then Placebo Stimulation: Participants first receive sub-threshold high-frequency spinal cord stimulation (1200 Hz frequency, 200 μsec pulse width, and an amplitude 90% of the threshold for detection of a sensory percept) for 2 weeks. After a 2-week washout period, they then received sham spinal cord stimulation (1200 Hz at 0 V amplitude) for 2 weeks."
- Total: Total of all reporting groups
Arm/Group | High-Frequency Stimulation, Then Placebo Stimulation | Placebo Stimulation, Then High-Frequency Stimulation | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Pain Scale
Description: Assessment of overall degree of back and leg pain during each phase of stimulation (ie conventional baseline stimulation, high-density stimulation, conventional "washout" stimulation, and sham stimulation). Scores range from 0 - 100, with a higher score indicating more pain.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- High-density Stimulation: All patients will receive 2 weeks of conventional spinal cord stimulation as a baseline (60 Hz, 200 usec, at an amplitude above sensory perception). Patients will then be randomly assigned to receive sub-threshold, high-density spinal cord stimulation (1200 Hz, 200 usec, at an amplitude of 90% of the sensory threshold) for 2 weeks. Patients will then get another 2 weeks of conventional stimulation as a "washout" period. Finally, they will get 2 weeks of sham stimulation (1200 Hz, 200 usec, 0 amplitude).
- Placebo Stimulation: All patients will receive 2 weeks of conventional spinal cord stimulation as a baseline (60 Hz, 200 usec, at an amplitude above sensory perception). Patients will then be randomly assigned to receive 2 weeks of sham stimulation (1200 Hz, 200 usec, 0 amplitude). Patients will then get another 2 weeks of conventional stimulation as a "washout" period. Finally, they will get 2 weeks of sub-threshold, high-density spinal cord stimulation (1200 Hz, 200 usec, at an amplitude of 90% of the sensory threshold) for 2 weeks.
Arm/Group | High-density Stimulation | Placebo Stimulation
Number analyzed (Participants) | 4 | 4
units on a scale | 2.29 (0.41) | 6.31 (1.22)

2. Secondary Outcome: Change in Brief Pain Inventory (BPI)
Description: The BPI assesses pain at its "worst," "least," "average," and "now" (current pain). Each item is rated on a scale of 0 - 10 with 10 indicating higher levels of pain. For purposes of this outcome measure, we focused on "now" (current pain)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-density Stimulation | Placebo Stimulation
Number analyzed (Participants) | 4 | 4
units on a scale | -2.0625 (1.21875) | 1.21875 (1.555819)

3. Secondary Outcome: Change in SF-36
Description: The SF-36 is a measure of quality of life, with scores ranging from 0 - 100, with higher scores indicating a higher quality of life.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-density Stimulation | Placebo Stimulation
Number analyzed (Participants) | 4 | 4
units on a scale | -28.125 (19.83001) | 23.125 (35.90352)

4. Secondary Outcome: Pain Vigilance and Awareness Questionnaire (PVAQ)
Description: The PVAQ is a measure of vigilance and attention to pain. Total scores can range from 0 to 90, with higher scores indicating more pain vigilance.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Stimulation: All patients will receive 2 weeks of conventional All patients will receive 2 weeks of conventional spinal cord stimulation as a baseline (60 Hz, 200 usec, at an amplitude above sensory perception). Patients will then be randomly assigned to receive 2 weeks of sham stimulation (1200 Hz, 200 usec, 0 amplitude). Patients will then get another 2 weeks of conventional stimulation as a "washout" period. Finally, they will get 2 weeks of sub-threshold, high-density spinal cord stimulation (1200 Hz, 200 usec, at an amplitude of 90% of the sensory threshold) for 2 weeks.
Arm/Group | High-density Stimulation | Placebo Stimulation
Number analyzed (Participants) | 4 | 4
units on a scale | 46.8 (7.1) | 51.5 (6.4)

5. Secondary Outcome: Number of Patients With Side Effects of Stimulation
Description: Incidence of side effects of stimulation
Time Frame: 8 weeks
Population: No subjects were randomized to the conventional spinal cord stimulation group
Measure: Number; unit: participants
Arm/Group | High-density Stimulation | Placebo Stimulation
Number analyzed (Participants) | 4 | 4
participants | 2 | 2

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: No subjects were enrolled in to the Conventional Spinal Cord Stimulation group
Groups:
- High-Frequency Stimulation: Participants received sub-threshold high-frequency spinal cord stimulation (1200 Hz frequency, 200 μsec pulse width, and an amplitude 90% of the threshold for detection of a sensory percept) for 2 weeks.
- Placebo Stimulation: Participants received sham spinal cord stimulation (1200 Hz at 0 V amplitude) for 2 weeks.
Arm/Group | High-Frequency Stimulation | Placebo Stimulation
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Frequency Stimulation (N=4) | Placebo Stimulation (N=4)
Paresthesia (Nervous system disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No